CLINICAL TRIAL: NCT02973633
Title: Diffusion MRI in Heart Failure
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David E Sosnovik, Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016P001898
Record Dates: First submitted 2016-11-19; First posted 2016-11-25 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Myocardial Infarction; Left Ventricular Hypertrophy
Keywords: Heart Failure; Remodeling; Myocardial Infarction; Left Ventricular Hypertrophy; Diffusion Tensor MRI
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Hypertrophy, Left Ventricular | interventions — Diffusion Tensor Imaging; gadolinium DOTA meglumine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Healthy Volunteers (Active Comparator): DTI will be performed in healthy volunteers to characterize normal fiber architecture in the heart and provide a comparison group for the patients imaged in the other arms.
  Interventions: Device: Diffusion Tensor MRI (DTI)
- Patients with Recent Myocardial Infarction (Active Comparator): Patients with recent ST elevation myocardial infarcts will be recruited and imaged serially with DTI to detect changes in fiber architecture and their correlation with remodeling of the left ventricle.
  Interventions: Device: Diffusion Tensor MRI (DTI); Drug: Gadolinium DOTA Meglumine
- Patients with Left Ventricular Hypertrophy (Active Comparator): Patients with left ventricular hypertrophy and a history of heart failure will be recruited and imaged serially with DTI to detect changes in fiber architecture and their correlation with the onset and progression of heart failure.
  Interventions: Device: Diffusion Tensor MRI (DTI)

INTERVENTIONS:
Device: Diffusion Tensor MRI (DTI) — Diffusion Tensor MRI (DTI) measures the diffusion of water in the heart, which allows the orientation of the muscle fibers in the heart to be determined.
Drug: Gadolinium DOTA Meglumine — Late Gadolinium enhancement
  Arms: Patients with Recent Myocardial Infarction

SUMMARY:
The development of symptomatic heart failure is frequently preceded by a pre-clinical period of structural remodeling in the heart. The remodeling process driving this transition, however, remains poorly understood. The investigators hypothesize that imaging the diffusion of water in the heart with MRI will allow its microstructure to be resolved. The investigators further hypothesize that the characterization of microstructural changes in the heart will help elucidate the pathogenesis of heart failure and the transition from a compensated to a decompensated state. Patients with recent myocardial infarcts and left ventricular hypertrophy, who are at risk for the development of heart failure, will be enrolled. The participants will undergo serial diffusion tensor MRI (DTI) imaging of the heart to characterize changes in myocardial microstructure over time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with no history of hypertension, diabetes or heart disease
* Patients with ST Elevation MI within last 6-10 weeks who are angina free, and have been seen by a cardiologist since discharge
* Patients with episode of heart failure within last 12 months and left ventricular hypertrophy, documented by echocardiogram or MRI.

Exclusion Criteria:

1. Presence of metallic foreign bodies/objects
2. Selected medical devices and implants
3. Pacemakers, implantable defibrillators, life vests
4. Coronary artery stent within last 6 weeks (unless the stent is a MRI-inert chromium-cobalt stent)
5. Known untreated ventricular arrhythmia such as sustained ventricular tachycardia within last 12 months
6. Atrial fibrillation that is not well rate controlled (heart rate >125)
7. Unstable angina within last 2 months that has not been fully evaluated by a cardiologist
8. Syncope within last 6 weeks
9. Hemodynamic instability (Systolic BP less than 100 or greater than 180)
10. Decompensated heart failure (inability to lie flat and perform a breath-hold).
11. Glomerular filtration rate (GFR) < 60 for those receiving gadolinium.
12. Labile GFR that is not stable/similar on last 2 measurements (for those receiving gadolinium).
13. Patients with GFR < 20 or on any form of dialysis.
14. Infiltrative cardiomyopathy (amyloid, sarcoid, hemachromatosis)
15. Recent surgery (within the last 3 months)
16. Prior stroke with large residual deficit
17. Presence of liver or respiratory failure
18. Pregnancy and nursing mothers
19. Claustrophobia
20. Known seizure disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Myofiber Helix Angle | 12 months
  The investigators aim to determine how the myofibers in the heart change their orientation in heart disease by measuring their helix angle.

SECONDARY OUTCOMES:
Correlation of Myofiber Helix Angle and Strain | 12 months
  The investigators aim to correlate how changes in fiber architecture correlate with changes in left ventricular strain.

CONTACTS AND LOCATIONS:
Overall Officials: David E. Sosnovik, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Result] Mekkaoui C, Reese TG, Jackowski MP, Cauley SF, Setsompop K, Bhat H, Sosnovik DE. Diffusion Tractography of the Entire Left Ventricle by Using Free-breathing Accelerated Simultaneous Multisection Imaging. Radiology. 2017 Mar;282(3):850-856. doi: 10.1148/radiol.2016152613. Epub 2016 Sep 28. PMID 27681278